CLINICAL TRIAL: NCT01015846
Title: Assessment of Transverse Abdominis Muscle Function Associated With Stabilization Exercises in Low Back Pain Patients
Brief Title: Ultrasound Assessment During Exercise
Acronym: Redcord RUSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Susan Saliba, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14046
Record Dates: First submitted 2009-09-28; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Low Back Pain
Keywords: Core; Redcord; RUSI; low back
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Exercise
- Core stability exercise (Active Comparator): Traditional core stability exercise
  Interventions: Other: Core stability exercise

INTERVENTIONS:
Other: Exercise — Redcord (sling exercise) and traditional exercise
  Arms: Intervention
Other: Core stability exercise — Traditional core stability exercise
  Arms: Core stability exercise

SUMMARY:
This study evaluates the ability of the transverse abdominis (TrA) to contract during and after two different types of exercise - either sling based exercise or traditional core stability exercise. The TrA is measured by real time ultrasound imaging. The investigators hypothesized that the sling based exercise would activate the TrA to a greater degree and that there would be a greater activation after the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain with stabilization classification

Exclusion Criteria:

* Fractures, neurological condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
TrA activation ratio measured by RUSI | Pre - during - post exercise during a single day

CONTACTS AND LOCATIONS:
Overall Officials: Susan Saliba, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Grooms DR, Grindstaff TL, Croy T, Hart JM, Saliba SA. Clinimetric analysis of pressure biofeedback and transversus abdominis function in individuals with stabilization classification low back pain. J Orthop Sports Phys Ther. 2013 Mar;43(3):184-93. doi: 10.2519/jospt.2013.4397. Epub 2012 Nov 16. PMID 23160344